CLINICAL TRIAL: NCT02636530
Title: Effect of Two Exercise Programs on Bone Strength and Architecture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-1451
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ground Reaction Forces (Experimental): Participants will have an individualized exercise program that includes walking, jogging, stair climbing, and box jumping.
  Interventions: Behavioral: Ground Reaction Forces
- Joint Reaction Forces (Experimental): Participants will have an individualized exercise program that includes weight lifting and aerobic rowing.
  Interventions: Behavioral: Joint Reaction Forces

INTERVENTIONS:
Behavioral: Ground Reaction Forces — 6 month exercise program that loads the body via gravitational forces.
  Arms: Ground Reaction Forces
Behavioral: Joint Reaction Forces — 6 month exercise program that loads the body via loading the joints.
  Arms: Joint Reaction Forces

SUMMARY:
Bone responds according to the load placed on it. In this study, investigators want to know if exercise that loads the body in exercises, like walking or jogging (Ground Reaction Forces: GRF), affects bone differently than exercises that load the joints, like weight lifting (Joint Reaction Forces: JRF). Participants will exercise at least 3 times a week for 6 months. Measures of bone strength and mass, muscular strength, and aerobic fitness will be taken at the beginning and the end of the 6 month program. Period blood samples will be taken for future analysis of blood markers.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* in generally good health
* not physically active (less than 60 minutes of purposeful exercise/week)
* able to travel to the exercise facility a minimum of 3 times/week

Exclusion Criteria:

* use of glucocorticoids
* abnormal resting EKG
* angina and/or evidence of acute myocardial ischemia during a treadmill test
* resting blood pressure above 150 mmHg systolic of 90 mmHg diastolic
* anti-resorptive drug use in the last 2 years
* initiation of treatments that could impact bone metabolism (diuretics, hormones, bine anabolic agents) in the prior 6 months
* dual-energy x-ray absorptiometry (DXA) t-score <+ -2.5 at the femoral neck and/or lumbar spine
* serum vitamin D concentration <20 ng/mL
* uncontrolled thyroid disease
* any contraindications to regular exercise

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Volumetric Bone Mineral Density (vBMD) | Baseline and 6 month
  Measured via quantitative computed tomography (QCT)
Change in Areal Bone Mineral Density (aBMD) | Baseline and 6 month
  Measured via dual-energy x-ray absorptiometry (DXA)
Change in Bone Strength | Baseline and 6 month
  Measured via finite element analysis (FEA) from QCT

SECONDARY OUTCOMES:
Change in 1-Repetition Maximum (1RM) | Baseline and 6 month
Change in Maximal Oxygen Uptake (cardiovascular fitness) | Baseline and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Veteran's Affairs Eastern Colorado Healthcare System, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No